CLINICAL TRIAL: NCT02028455
Title: Pediatric and Young Adult Leukemia Adoptive Therapy (PLAT)-02: A Phase 1/2 Feasibility and Safety Study of CD19-CAR T Cell Immunotherapy for CD19+ Leukemia
Brief Title: A Pediatric and Young Adult Trial of Genetically Modified T Cells Directed Against CD19 for Relapsed/Refractory CD19+ Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLAT-02
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: CD19+ Acute Leukemia
Keywords: pediatric; young adult; acute lymphoblastic leukemia; CD19; leukemia; Chimeric Antigen Receptor; T cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1 - Cohort 1A (Experimental): This phase 1 cohort will receive Patient Derived CD19 specific CAR T cells at a dose of 5x10^5 CAR T cells/kg
  Interventions: Biological: Patient Derived CD19 specific CAR T cells also expressing an EGFRt
- Phase 1 - Cohort 1B (Experimental): This phase 1 cohort will receive Patient Derived CD19 specific CAR T cells at a dose of 1x10^6 CAR T cells/kg
  Interventions: Biological: Patient Derived CD19 specific CAR T cells also expressing an EGFRt
- Phase 1 - Cohort 1C (Experimental): This phase 1 cohort will receive Patient Derived CD19 specific CAR T cells at a dose of 5x10^6 CAR T cells/kg
  Interventions: Biological: Patient Derived CD19 specific CAR T cells also expressing an EGFRt
- Phase 1 - Cohort 1D (Experimental): This phase 1 cohort will receive Patient Derived CD19 specific CAR T cells at a dose of 1x10^7 CAR T cells/kg
  Interventions: Biological: Patient Derived CD19 specific CAR T cells also expressing an EGFRt
- Phase 1 - Cohort 1F1 (Experimental): This phase 1 cohort will receive Patient Derived CD19 specific CAR T cells at a dose of 5x10^5 CAR T cells/kg following prescribed lymph-depletion with fludarabine and cyclophosphamide
  Interventions: Biological: Patient Derived CD19 specific CAR T cells also expressing an EGFRt
- Phase 1 - Cohort 1F2 (Experimental): This phase 1 cohort will receive Patient Derived CD19 specific CAR T cells at a dose of 1x10^6 CAR T cells/kg following prescribed lymph-depletion with fludarabine and cyclophosphamide
  Interventions: Biological: Patient Derived CD19 specific CAR T cells also expressing an EGFRt
- Phase 2 (Experimental): The phase 2 cohort will receive Patient Derived CD19 specific CAR T cells at a dose of 1 x 10^6 CAR T cells/kg following lymphodepletion if indicated.
  Interventions: Biological: Patient Derived CD19 specific CAR T cells also expressing an EGFRt

INTERVENTIONS:
Biological: Patient Derived CD19 specific CAR T cells also expressing an EGFRt — Defined Composition CD4 and CD8 T cells Lentivirally Transduced to Express a Second Generation 4-1BB:zeta CD19 CAR and EGFRt

SUMMARY:
Patients with relapsed or refractory leukemia often develop resistance to chemotherapy. For this reason, we are attempting to use T cells obtained directly from the patient, which can be genetically modified to express a chimeric antigen receptor (CAR). The CAR enables the T cell to recognize and kill the leukemic cell through the recognition of CD19, a protein expressed of the surface of the leukemic cell in patients with CD19+ leukemia. This is a phase 1/2 study designed to determine the maximum tolerated dose of the CAR+ T cells as well as to determine the efficacy. The phase 1 cohort is restricted to those patients who have already had an allogeneic hematopoietic cell transplant (HCT). The phase 2 is open to all patients regardless of having a history of HCT.

DETAILED DESCRIPTION:
Upon meeting the eligibility requirements and enrolling on study, subjects will undergo apheresis to obtain the T cells for the generation of the CD19 CAR+ T cells. In patients with a prior history of allogeneic HCT, the T cells obtained are of donor origin. The T cells are isolated from the apheresis product, the CD4 and CD8 T cells are then selected and grown separately, transduced with a lentivirus to express the CD19 CAR as well as a truncated EGFR that has no signaling capacity (noted EGFRt) and expanded in culture over a three week period. During the process of cell generation, subjects will continue to be cared for by their primary oncologist and may undergo additional treatment directed at the leukemia during this time.

After the CAR+ T cells have been generated, the subject undergoes a disease assessment and determination if lymphodepletion is necessary. A variety of lymphodepletion strategies are acceptable and determined on a case by case basis. At least 48 hours after the completion of lymphodepletion, the subject will receive and infusion of CAR+ T cells at an approximate 1:1 ratio of CD4 to CD8 CAR+ T cells.

Following treatment with the CAR+ T cells, subjects will be followed intensely for 2 months with serial blood testing and re-evaluation of disease status with bone marrow aspirates. After 2 months, the subjects clinical care will be resumed by their primary oncologist, and it is possible that they would receive additional chemotherapy or HCT.

Some subjects will receive cetuximab for ablation of the genetically modified T cells. Criteria to receive cetuximab include acute toxicities that are life threatening, as well as an ongoing remission with continued B cell aplasia.

Upon completion of the study, subjects will be followed bi-annually for 5 years, and then annually for 10 additional years with either a medical history, physical exam and blood tests or a phone call/questionnaire. This follow up will help to determine if the subject develops any long-term health problems related to the CAR+ T cells including a new cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients must be ≥12 months of age and <27 years of age at the time of study enrollment.

Must be ≥10kg

Confirmed CD19+ leukemia recurrence defined as ≥0.01% disease in the marrow or isolated extramedullary disease following allogeneic HCT. [N.B. Study closed to enrollment of leukemia subjects]

OR

No prior history of allogeneic HCT (one of the following)

* 2nd or greater relapse, with or without extramedullary disease (isolated extramedullary disease is eligible)
* 1st marrow relapse at end of 1st month of re-induction with marrow having ≥0.01% blast disease, with or without extramedullary disease
* Primary Refractory as defined as having M2 or M3 marrow after induction
* Subject has indication for HCT but has been deemed ineligible

OR

CD19+ Non-Hodgkin Lymphoma (NHL) refractory or relapsed with no known curative therapies available [N.B. Study remains open to enrollment of lymphoma subjects]

Patients with CNS involvement are eligible provided that they are asymptomatic and in the opinion of the study PI have a reasonable expectation that disease burden can be controlled in the interval between enrollment and T cell infusion. Patients that have a significant neurologic deterioration will be not be eligible for T cell infusion until alternate therapies result in neurological stabilization.

Patients must have a Lansky performance status score of ≥50 or a Karnofsky score of ≥ 50 for patients ≥16 years of age.

Life Expectancy of >8 weeks

Patients must be free from active GVHD and off immunosuppressive GVHD therapy for 4 weeks prior to enrollment.

Recovered from acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy

It must be at least 7 days since last chemotherapy was administered (this does not include intrathecal chemotherapy or maintenance chemotherapy)

No systemic corticosteroids (unless physiologic replacement dosing) within 7 days of enrollment.

No prior genetically modified cell therapy that is still detectable or virotherapy allowed.

* Normal serum creatinine based on age/gender
* Total bilirubin </3x ULN OR conjugated bilirubin </2mg/dl
* ALT </5X ULN
* SF of >28% by ECHO or EF >50% by MUGA
* ALC of >/= 100 cells/ul
* Pulse ox >/= 90% on room air

Patient must have documented negative HIV antigen and antibody, Hepatitis B surface antigen, and Hepatitis C antibody within 3 months prior to enrollment. For patient with positive Hepatitis C Ab, negative PCR testing must be documented in order to be eligible.

Patients must NOT have active clinically significant CNS dysfunction (including but not limited to such as uncontrolled seizure disorder, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder)

Must agree to highly effective contraception during and for 12 months after T cell infusion.

Patients must be able to tolerate apheresis procedure, including placement of temporary apheresis line if required.

Patients must NOT have an active malignancy other than CD19+ leukemia.

Patients must NOT have an active severe infection defined as:

* A positive blood culture within 48 hours of study enrollment
* A fever above 38.2 C AND clinical signs of infection within 48 hours of study enrollment

Patients must NOT have any concurrent medical condition that, in the opinion of the PI or designee, would prevent the patient from undergoing protocol-based therapy. Patients with a primary immunodeficiency/ bone marrow failure syndrome are excluded from this trial.

Research participant or parent/legal guardian must agree to participate in long-term follow-up for up to 15 years, if they are enrolled in the study and receive T-cell infusion.

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 167 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2036-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Annesley, MD, Study Chair — Seattle Children's Hospital
Locations (3):
- United States (3):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Oakland, Oakland, California
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Annesley C, Seidel K, Wu Q, Summers C, Wayne AS, Pulsipher MA, Agrawal AK, Brown CT, Mgebroff S, Lindgren C, Rawlings-Rhea S, Huang W, Wilson AL, Jensen MC, Park JR, Gardner RA. Outcomes of PLAT-02 and PLAT-03: evaluating CD19 CAR T-cell therapy and CD19-expressing T-APC support in pediatric B-ALL. Blood. 2025 Aug 14;146(7):789-801. doi: 10.1182/blood.2025028359. PMID 40233328
- [Derived] Ceppi F, Wilson AL, Annesley C, Kimmerly GR, Summers C, Brand A, Seidel K, Wu QV, Beebe A, Brown C, Mgebroff S, Lindgren C, Rawlings-Rhea SD, Huang W, Pulsipher MA, Wayne AS, Park JR, Jensen MC, Gardner RA. Modified Manufacturing Process Modulates CD19CAR T-cell Engraftment Fitness and Leukemia-Free Survival in Pediatric and Young Adult Subjects. Cancer Immunol Res. 2022 Jul 1;10(7):856-870. doi: 10.1158/2326-6066.CIR-21-0501. PMID 35580141
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Finney OC, Brakke HM, Rawlings-Rhea S, Hicks R, Doolittle D, Lopez M, Futrell RB, Orentas RJ, Li D, Gardner RA, Jensen MC. CD19 CAR T cell product and disease attributes predict leukemia remission durability. J Clin Invest. 2019 Mar 12;129(5):2123-2132. doi: 10.1172/JCI125423. Print 2019 May 1. PMID 30860496
- [Derived] Gardner RA, Finney O, Annesley C, Brakke H, Summers C, Leger K, Bleakley M, Brown C, Mgebroff S, Kelly-Spratt KS, Hoglund V, Lindgren C, Oron AP, Li D, Riddell SR, Park JR, Jensen MC. Intent-to-treat leukemia remission by CD19 CAR T cells of defined formulation and dose in children and young adults. Blood. 2017 Jun 22;129(25):3322-3331. doi: 10.1182/blood-2017-02-769208. Epub 2017 Apr 13. PMID 28408462
- [Derived] Gardner R, Wu D, Cherian S, Fang M, Hanafi LA, Finney O, Smithers H, Jensen MC, Riddell SR, Maloney DG, Turtle CJ. Acquisition of a CD19-negative myeloid phenotype allows immune escape of MLL-rearranged B-ALL from CD19 CAR-T-cell therapy. Blood. 2016 May 19;127(20):2406-10. doi: 10.1182/blood-2015-08-665547. Epub 2016 Feb 23. PMID 26907630

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 - Cohort 1A: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 5x10^5 CAR T cells/kg
- Phase 1 - Cohort 1B: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 1x10^6 CAR T cells/kg
- Phase 1 - Cohort 1C: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 5x10^6 CAR T cells/kg
- Phase 1 - Cohort 1D: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 1x10^7 CAR T cells/kg
- Phase 1 - Cohort 1F1: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 5x10^5 CAR T cells/kg following prescribed lymphodepletion with fludarabine and cyclophosphamide
- Phase 1 - Cohort 1F2: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 1x10^6 CAR T cells/kg following prescribed lymphodepletion with fludarabine and cyclophosphamide
- Phase 1- Not Treated: Phase 1 subjects who were not treated
- Phase 2: The phase 2 cohort received Patient Derived CD19 specific CAR T cells at a dose of 1 x 10^6 CAR T cells/kg following lymphodepletion if indicated.
Period: Enrollment and Preliminary Assessments
Arm/Group | Phase 1 - Cohort 1A | Phase 1 - Cohort 1B | Phase 1 - Cohort 1C | Phase 1 - Cohort 1D | Phase 1 - Cohort 1F1 | Phase 1 - Cohort 1F2 | Phase 1- Not Treated | Phase 2
Started | 7 | 12 | 7 | 5 | 6 | 6 | 4 | 120
Completed | 7 | 12 | 7 | 5 | 6 | 6 | 0 | 103
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 17
Not completed — Went off study without receiving CAR T cell infusion | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 17
Period: Treatment(T Cell Infusion) and Follow up
Arm/Group | Phase 1 - Cohort 1A | Phase 1 - Cohort 1B | Phase 1 - Cohort 1C | Phase 1 - Cohort 1D | Phase 1 - Cohort 1F1 | Phase 1 - Cohort 1F2 | Phase 1- Not Treated | Phase 2
Started | 7 | 12 | 7 | 5 | 6 | 6 | 0 | 103
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 12 | 7 | 5 | 6 | 6 | 0 | 103
Not completed — Death | 4 | 9 | 3 | 5 | 3 | 2 | 0 | 40
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Still in long-term follow up | 3 | 3 | 4 | 0 | 3 | 3 | 0 | 61

BASELINE CHARACTERISTICS:
Groups:
- Phase 1-Cohort 1A: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 5x10^5 CAR T cells/kg
- Phase 1-Cohort 1B: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 1x10^6 CAR T cells/kg
- Phase 1-Cohort 1C: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 5x10^6 CAR T cells/kg
- Phase 1-Cohort 1D: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 1x10^7 CAR T cells/kg
- Phase 1-Cohort 1F1: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 5x10^5 CAR T cells/kg following prescribed lymphodepletion with fludarabine and cyclophosphamide
- Phase 1-Cohort 1F2: This phase 1 cohort received Patient Derived CD19 specific CAR T cells at a dose of 1x10^6 CAR T cells/kg following prescribed lymphodepletion with fludarabine and cyclophosphamide
- Phase 1 - Not Treated: This phase 1 cohort did not receive Patient Derived CD19 specific CAR T cells
- Phase 2: The phase 2 cohort received Patient Derived CD19 specific CAR T cells following lymphodepletion if indicated
- Total: Total of all reporting groups
Arm/Group | Phase 1-Cohort 1A | Phase 1-Cohort 1B | Phase 1-Cohort 1C | Phase 1-Cohort 1D | Phase 1-Cohort 1F1 | Phase 1-Cohort 1F2 | Phase 1 - Not Treated | Phase 2 | Total
Number analyzed (Participants) | 7 | 12 | 7 | 5 | 6 | 6 | 4 | 120 | 167
Age, Continuous [Median (Full Range); unit: years] | 19 [5 to 22] | 9 [1 to 23] | 15 [2 to 20] | 6 [1 to 22] | 10 [1 to 25] | 13.5 [4 to 21] | 11 [8 to 14] | 13 [1 to 26] | 13 [1 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 5 | 3 | 4 | 1 | 40 | 63
  Male | 3 | 9 | 4 | 0 | 3 | 2 | 3 | 80 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 2 | 2 | 0 | 1 | 1 | 38 | 49
  Not Hispanic or Latino | 6 | 8 | 5 | 3 | 5 | 4 | 2 | 72 | 105
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 10 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 5
  White | 5 | 8 | 4 | 2 | 5 | 3 | 3 | 66 | 96
  More than one race | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 6
  Unknown or Not Reported | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 39 | 49
Diagnosis [Count of Participants; unit: Participants]
  Leukemia | 7 | 12 | 7 | 5 | 6 | 6 | 4 | 106 | 153
  Non Hodgkin's Lymphoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event Meeting the Dose-Limiting Toxicity Definition
Description: The safety of the T cell infusion at the maximum tolerated dose determined in Phase 1, and further characterized in Phase 2, will be described
Time Frame: Initial CAR T cell infusion through 30 days post infusion
Population: Phase 1 cohorts: Toxicity-evaluable leukemia patients who received CAR T cells; Phase 2 cohort: Toxicity-evaluable leukemia patients treated with the Phase 2 dose, 1 x 10^6 CAR T cells/kg, following lymphodepletion with fludarabine and cyclophosphamide
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Cohort 1A | Phase 1-Cohort 1B | Phase 1-Cohort 1C | Phase 1-Cohort 1D | Phase 1-Cohort 1F1 | Phase 1-Cohort 1F2 | Phase 2
Number analyzed (Participants) | 7 | 12 | 7 | 5 | 6 | 6 | 81
Participants
  Number of participants who experienced an AE meeting the Dose-Limiting Toxicity definition | 1 | 1 | 2 | 2 | 0 | 1 | 17
  Number of participants who did not experience an AE meeting the Dose-Limiting Toxicity definition | 6 | 11 | 5 | 3 | 6 | 5 | 64

2. Primary Outcome: Number of Participants With an MRD Negative Complete Remission After Initial CAR T Cell Infusion
Description: The efficacy of the T cell infusion will be estimated based on the number of participants who have an MRD negative bone marrow aspirate following the initial T cell infusion
Time Frame: Initial CAR T cell infusion through Day 63 post infusion assessment (+/- 14 days)
Population: Efficacy-evaluable leukemia patients in Phase 2, plus Phase 1 patients treated at the Phase 2 dose in cohort 1F2, who received SCRIv1 or SCRIv1.5 CAR T cells following prescribed lymphodepletion with fludarabine and cyclophosphamide
Measure: Count of Participants; unit: Participants
Groups:
- SCRI-CAR19v1/v1.5 Efficacy-evaluable Leukemia Cohort: Efficacy-evaluable leukemia patients who received SCRIv1 or SCRIv1.5 CAR T cells
Arm/Group | SCRI-CAR19v1/v1.5 Efficacy-evaluable Leukemia Cohort
Number analyzed (Participants) | 71
Participants
  Number of Participants with an MRD Negative Complete Remission after Initial CAR T Infusion | 63
  Number of Participants without an MRD Negative Complete Remission after Initial CAR T Infusion | 8

3. Primary Outcome: Number of Participants Who Have a Releasable Cell Product Generated
Description: The feasibility of manufacturing and releasing T cell products from pediatric and young adult patients with CD19+ relapsed or refractory leukemia
Time Frame: Up to 28 days per manufacturing attempt
Population: Participants evaluable for manufacturing feasibility.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: The phase 2 cohort received Patient Derived CD19 specific CAR T cells at a dose of 1x10^6 CAR T cells/kg following lymphodepletion if indicated
Arm/Group | Phase 1-Cohort 1A | Phase 1-Cohort 1B | Phase 1-Cohort 1C | Phase 1-Cohort 1D | Phase 1-Cohort 1F1 | Phase 1-Cohort 1F2 | Phase 1 - Not Treated | Phase 2
Number analyzed (Participants) | 7 | 12 | 7 | 5 | 6 | 6 | 3 | 119
Participants
  Number of participants for whom a releasable CAR T cell product was manufactured | 7 | 12 | 7 | 5 | 6 | 6 | 1 | 116
  Number of participants for whom no releasable CAR T cell product was manufactured | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3

4. Secondary Outcome: Persistence of Functional CD19 CAR+ T Cells
Description: Participants will be followed for 63 days to determine if the transferred T cells remain detectable in the blood and bone marrow
Time Frame: Initial CAR T Infusion through Day 63 post infusion assessment (+/- 14 days)
Population: Efficacy-evaluable leukemia patients in Phase 2, plus Phase 1 patients treated at the Phase 2 dose in Cohort 1F2, who received SCRIv1 or SCRIv1.5 CAR T cells following prescribed lymphodepletion with fludarabine and cyclophosphamide and who were followed for loss of persistence through the Day 63 assessment window. Excludes one participant with insufficient samples collected to determine Day 63 persistence status.
Measure: Count of Participants; unit: Participants
Groups:
- SCRI-CAR19v1/v1.5 Efficacy- and Persistence-evaluable Leukemia Cohort: Participants from the efficacy-evaluable leukemia population who were followed for loss of persistence through the d63 assessment window.
Arm/Group | SCRI-CAR19v1/v1.5 Efficacy- and Persistence-evaluable Leukemia Cohort
Number analyzed (Participants) | 70
Participants
  Number of participants with functional CAR T cell persistence through the Day 63 study assessment | 42
  Number of participants without functional CAR T cell persistence through the Day 63 study assessment | 28

5. Secondary Outcome: Number of Participants With Recrudescence or Development of Acute GVHD (Graft Versus Host Disease) Symptoms Post CAR T Infusion
Time Frame: Initial CAR T Infusion through Day 63 post infusion assessment (+/- 14 days)
Population: Number of participants with a history of prior allogeneic HSCT (hematopoietic stem cell transplantation) who received CAR T infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Cohort 1A | Phase 1-Cohort 1B | Phase 1-Cohort 1C | Phase 1-Cohort 1D | Phase 1-Cohort 1F1 | Phase 1-Cohort 1F2 | Phase 2
Number analyzed (Participants) | 7 | 7 | 4 | 3 | 4 | 3 | 36
Participants
  Number of subjects without recrudescence or development of Acute GVHD symptoms post CAR T infusion | 6 | 7 | 4 | 3 | 4 | 3 | 36
  Number of subjects with recrudescence or development of Acute GVHD symptoms post CAR T infusion | 1 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants That Received Cetuximab Who Have T Cells Successfully Ablated
Description: The efficacy of cetuximab to ablate the T cells will be measured by loss of detection of T cells and any associated toxicities as well as facilitating B cell recovery.
Time Frame: 3 years
Population: Number of subjects receiving cetuximab on study for ablation of CAR T cells
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Cohort 1A | Phase 1-Cohort 1B | Phase 1-Cohort 1C | Phase 1-Cohort 1D | Phase 1-Cohort 1F1 | Phase 1-Cohort 1F2 | Phase 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Participants
  Number of participants receiving cetuximab on study for ablation of CAR T cells | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Number of participants whose CAR T cells were successfully ablated by cetuximab administration | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse event data are systematically collected from initiation of infusion through 30 days post CAR T infusion. Serious Adverse Event reports with an attribution of Possibly, Probably or Definitely related to CAR T cells are included in the data up to 1 year post-infusion.
Description: Adverse events were assessed using NCI Common Terminology Criteria for Adverse Events v4.0, except for Cytokine Release Syndrome during Phase 2, which was assessed using modified Lee criteria.* Neurotoxicity and CRS events with grade >=1 and other events with grade >=2 were systematically captured
  *Lee DW, Gardner R, Porter DL, Louis CU, Ahmed N, Jensen M, Grupp SA, Mackall CL. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014 Jul 10;124(2):188-95.
Groups:
- Phase 1 - Cohort 1F1: This phase 1 cohort will receive Patient Derived CD19 specific CAR T cells at a dose of 5x10^5 CAR T cells/kg following prescribed lymphodepletion with fludarabine and cyclophosphamide
- Phase 1 - Cohort 1F2: This phase 1 cohort will receive Patient Derived CD19 specific CAR T cells at a dose of 1x10^6 CAR T cells/kg following prescribed lymphodepletion with fludarabine and cyclophosphamide
Arm/Group | Phase 1 - Cohort 1A | Phase 1 - Cohort 1B | Phase 1 - Cohort 1C | Phase 1 - Cohort 1D | Phase 1 - Cohort 1F1 | Phase 1 - Cohort 1F2 | Phase 2
All-Cause Mortality (participants affected / at risk) | 4/7 | 9/12 | 3/7 | 5/5 | 3/6 | 2/6 | 40/103
Serious Adverse Events (participants affected / at risk) | 6/7 | 10/12 | 5/7 | 5/5 | 2/6 | 4/6 | 48/103
Other Adverse Events (participants affected / at risk) | 7/7 | 12/12 | 7/7 | 5/5 | 6/6 | 6/6 | 103/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Cohort 1A (N=7) | Phase 1 - Cohort 1B (N=12) | Phase 1 - Cohort 1C (N=7) | Phase 1 - Cohort 1D (N=5) | Phase 1 - Cohort 1F1 (N=6) | Phase 1 - Cohort 1F2 (N=6) | Phase 2 (N=103)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Heart Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial Tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Optic Nerve Disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3
Anaphylaxis (Immune system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Cytokine Release Syndrome (Immune system disorders) | 2 | 5 | 5 | 3 | 1 | 3 | 22
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter Related Infection (Infections and infestations) | 0 | 4 | 0 | 3 | 1 | 1 | 0
Gram-Positive Bacterial Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Periorbital Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Skin Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Yeast Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Creatinine Increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaw Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Progressive Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Edema Cerebral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 4 | 3 | 3 | 0 | 2 | 12
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Intracranial Hemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 7
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3
Laryngeal Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Capillary Leak Syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Cohort 1A (N=7) | Phase 1 - Cohort 1B (N=12) | Phase 1 - Cohort 1C (N=7) | Phase 1 - Cohort 1D (N=5) | Phase 1 - Cohort 1F1 (N=6) | Phase 1 - Cohort 1F2 (N=6) | Phase 2 (N=103)
Anemia (Blood and lymphatic system disorders) | 4 | 11 | 6 | 4 | 5 | 3 | 60
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 8 | 4 | 2 | 5 | 2 | 15
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 | 10 | 6 | 1 | 5 | 4 | 36
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 3
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Optic Nerve Disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 8
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 0 | 2 | 1 | 0 | 8
Gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4 | 0 | 2 | 0 | 0 | 17
Oral Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Perirectal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 0 | 0 | 11
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2
Fever (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 6
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 10
Allergic Reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Cytokine Release Syndrome (Immune system disorders) | 4 | 7 | 1 | 2 | 5 | 2 | 68
Igg Decreased (Immune system disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 6
Catheter Related Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 5
Enterocolitis Infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 1
Mucosal Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 2
Nail Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 4
Upper Respiratory Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 4
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 12
Alanine Aminotransferase Increased (Investigations) | 2 | 2 | 2 | 0 | 1 | 0 | 10
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 8
Blood Bilirubin Increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 12
Creatinine Increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 2
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fibrinogen Decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 7
Lymphocyte Count Decreased (Investigations) | 2 | 5 | 3 | 1 | 0 | 0 | 20
Neutrophil Count Decreased (Investigations) | 5 | 7 | 6 | 3 | 4 | 5 | 55
Platelet Count Decreased (Investigations) | 5 | 8 | 4 | 4 | 4 | 1 | 42
Urine Output Decreased (Investigations) | 2 | 5 | 2 | 3 | 0 | 0 | 0
Weight Gain (Investigations) | 1 | 4 | 0 | 0 | 0 | 0 | 3
Weight Loss (Investigations) | 0 | 1 | 2 | 1 | 0 | 0 | 4
White Blood Cell Decreased (Investigations) | 5 | 8 | 6 | 1 | 3 | 4 | 46
Anorexia (Metabolism and nutrition disorders) | 1 | 6 | 0 | 0 | 1 | 1 | 13
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 6
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 7
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 2 | 1 | 1 | 9
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 6 | 2 | 4 | 1 | 1 | 11
Hypokalemia (Metabolism and nutrition disorders) | 2 | 4 | 2 | 4 | 1 | 1 | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 6 | 1 | 4 | 1 | 1 | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 4
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 5
Pain-Left Side (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 3
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 9
Headache (Nervous system disorders) | 5 | 2 | 3 | 1 | 1 | 3 | 32
Neuropathic Pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0 | 1 | 1 | 2 | 17
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 13
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomania (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 3
Nightmares (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polydipsia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 6
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal Diaper Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Skin GVHD (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Capillary Leak Syndrome (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 7 | 2 | 3 | 0 | 2 | 10
Hypotension (Vascular disorders) | 1 | 4 | 0 | 1 | 1 | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT02028455/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT02028455/SAP_001.pdf